CLINICAL TRIAL: NCT02412618
Title: A Randomized Comparison of Same-Day Oral Mifepristone-Misoprostol to Misoprostol Only for Cervical Preparation in Second Trimester Surgical Abortion
Brief Title: Same-Day Mifepristone-Misoprostol Compared to Misoprostol Only for Surgical Abortion Cervical Preparation
Acronym: MMSAP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medstar Health Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2012-245
Record Dates: First submitted 2015-03-13; First posted 2015-04-09 (Estimated); Results first posted 2022-03-02 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Induced Abortion
MeSH Terms: interventions — Mifepristone; Misoprostol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mifepristone (Active Comparator): Mifepristone 200mg oral tablet, once Misoprostol 400 mcg tablets, vaginally, once
  Interventions: Drug: Mifepristone; Drug: Misoprostol
- Placebo (Placebo Comparator): Placebo oral tablets, odorless, colorless and matched to Mifepristone appearance Misoprostol 400 mcg tablets, vaginally, once
  Interventions: Drug: Misoprostol; Dietary Supplement: Placebo

INTERVENTIONS:
Drug: Mifepristone — Progesterone antagonist
  Other Names: Mifeprex
  Arms: Mifepristone
Drug: Misoprostol — Prostaglandin E1
  Other Names: Cytotec
Dietary Supplement: Placebo — Tasteless, odorless, sugar based pill
  Arms: Placebo

SUMMARY:
A randomized double---blinded comparison of same---day mifepristone and misoprostol with misoprostol only for cervical preparation in second---trimester surgical abortion in 100 women at 14 0/7---19 6/7 weeks gestation.

DETAILED DESCRIPTION:
Women desiring abortion at gestational ages between 14 weeks 0 days and 19 weeks 6 days were randomized to 200-mg mifepristone or identical placebo with 400-mcg misoprostol vaginally 4-6 hours prior to D&E. Primary outcome was cervical dilation assessed by the largest Hegar dilator accepted without resistance. Secondary outcomes included total procedure time, and patient and provider perceptions. The study was powered to detect a 2-mm difference in cervical dilatation with 48 participants in each arm.

ELIGIBILITY:
Inclusion Criteria:

* healthy women
* eligible for non---urgent D&E
* 14 0/7 weeks to 19 6/7 weeks gestation, confirmed by sonogram

Exclusion Criteria:

* emergent need for D&E
* fetal demise
* intolerance
* allergy or contraindication to mifepristone or misoprostol

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2012-09; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

REFERENCES:
- [Derived] Casey FE, Ye PP, Perritt JD, Moreno-Ruiz NL, Reeves MF. A randomized controlled trial evaluating same-day mifepristone and misoprostol compared to misoprostol alone for cervical preparation prior to second-trimester surgical abortion. Contraception. 2016 Aug;94(2):127-33. doi: 10.1016/j.contraception.2016.02.032. Epub 2016 Mar 4. PMID 26948184

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Mifepristone | Placebo
Started | 50 | 50
Completed | 48 | 48
Not Completed | 2 | 2
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Expulsion | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mifepristone | Placebo | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 50 | 50 | 100
  >=65 years | 0 | 0 | 0
Sex/Gender, Customized [Number; unit: Participants]
  Female | 50 | 50 | 100

OUTCOME MEASURES:

1. Primary Outcome: Initial Cervical Dilation
Description: Initial cervical dilation as measured by Hegar Dilator accepted with least resistance
Time Frame: Assessed 4-6 hour following medications at time of D&E procedure
Measure: Mean (95% Confidence Interval); unit: mm
Arm/Group | Mifepristone | Placebo
Number analyzed (Participants) | 48 | 48
mm | 11.7 [9 to 13] | 10.9 [9 to 13]

2. Secondary Outcome: Patient Acceptability and Assessment of Pain and Side Effects (5-point Likert Scale)
Description: 5-point Likert scale given to patients following procedure once recovered from anesthesia assessing pain, side effects including nausea, vomiting, diarrhea, cramping, and if they would choose the method again or recommend to friends.
  Likert scale: Strongly agree (5), Agree (4), Neutral (3), Disagree (2), Strongly Disagree (1)
Time Frame: intraoperative
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Mifepristone | Placebo
Number analyzed (Participants) | 48 | 48
units on a scale
  Nausea | 4 [1 to 5] | 4 [1 to 5]
  Severe Cramps | 4 [1 to 5] | 4 [1 to 5]

ADVERSE EVENTS:
Arm/Group | Placebo | Mifepristone
All-Cause Mortality (participants affected / at risk) | 0/48 | 0/48
Serious Adverse Events (participants affected / at risk) | 0/48 | 0/48
Other Adverse Events (participants affected / at risk) | 0/48 | 0/48

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No